CLINICAL TRIAL: NCT03058341
Title: The Effect of Total Intravenous Anaesthesia With Propofol on Postoperative Pain After Third Molar Surgery: A Double-Blind Randomized Controlled Trial
Brief Title: Effect of Total Intravenous Anaesthesia With Propofol on Postoperative Pain After Bilateral Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW16-554
Record Dates: First submitted 2017-02-07; First posted 2017-02-20 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; propofol; TIVA
MeSH Terms: conditions — Pain, Postoperative | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Patients in the first group (S) will be anaesthetized by inhalational anaesthesia using sevoflurane. The patients in the second group (P) will be anaesthetized using total intravenous propofol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will not be informed about what type of anaesthesia they will receive. A separate investigator assessing the patients for data collection after the operation will be blinded. The anaesthetist providing general anaesthesia will not be involved in data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Sham Comparator): Patients will be anaesthetized by inhalational anaesthesia using sevoflurane.
  Interventions: Drug: Sevoflurane
- Group P (Experimental): Patients will be anaesthetized using total intravenous propofol.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — Monitoring and other anaesthetic procedures including the management of hypertension and hypotension will be the same as group S. The only difference is that induction and maintenance of general anaesthesia will be conducted using total intravenous infusion of propofol. Sevoflurane will not be used, and oxygen and air would be given to provide a FiO2 of 30-50%.
  Arms: Group P
Drug: Sevoflurane — Propofol 1.5-3mg/kg, remifentanil 0.5-1mcg/kg, and rocuronium 0.6-1mg/kg or atracurium 0.5mg/kg will be used intravenously (IV) for induction of general anaesthesia. Otrivin can be applied nasally at the discretion of the anaesthetist. Intubation would be performed after induction of general anaesthesia. General anaesthesia monitoring will be used. Sevoflurane, air and oxygen will be used for maintenance of general anaesthesia. FiO2 will be kept between 35-50%. BIS monitoring will be applied and level of anaesthetia will be titrated to keep a BIS value of 40-60. Intravenous remifentanil infusion between 0.1-0.25mcg/kg/min will be given and this will be titrated to optimal haemodynamic parameters. Muscle relaxants can be given during the operation as required.
  Arms: Group S

SUMMARY:
Propofol is one of the most commonly used intravenous anaesthetic drugs both for induction and maintenance of general anaesthesia. Some of the advantages of total intravenous anaesthesia (TIVA) with propofol include reduced nausea and vomiting, reduced atmospheric pollution, better wake up profile and a more favourable intracranial physiology. However, the need for a reliable intravenous access, specialized pumps, pain on injection and potential concerns regarding awareness are some reasons that preclude more common use.

Postoperative dental pain produces an inflammatory pain model. Since propofol has anti-inflammatory effects, it may have significant analgesic effects in patients undergoing dental surgery. To the best of our knowledge, there are no randomized controlled trials comparing the effects of TIVA propofol and inhalational anaesthetic on postoperative dental pain. The aim of this study is to investigate the effect of TIVA propofol on postoperative pain scores, analgesic consumption, and adverse effects in patients undergoing dental surgery. This will help determine whether propofol may be a useful analgesic adjunct in dental surgery.

DETAILED DESCRIPTION:
Preoperative care

Assessment will be done at the preadmission clinic or at the general ward. Fasting for patients will start at midnight before operation. Sedative premedication will not be prescribed.

Anaesthesia and intraoperative care

Group S

Patients from group S will be anaesthetized according to the following protocol:

On arrival to the operation theatre, a 20 or 22 gauge intravenous cannula will be inserted. Standard monitoring with pulse oximeter, non-invasive blood pressure, and three lead electrocardiogram will be applied prior to induction. Non-invasive blood pressure will be checked at least every 5 minutes throughout the operation.

Propofol 1.5-3mg/kg, remifentanil 0.5-1mcg/kg, and rocuronium 0.6-1mg/kg or atracurium 0.5mg/kg will be used intravenously (IV) for induction of general anaesthesia. Otrivin can be applied nasally at the discretion of the anaesthetist. Intubation would be performed after induction of general anaesthesia. General anaesthesia monitoring will be used. Sevoflurane, air and oxygen will be used for maintenance of general anaesthesia. FiO2 will be kept between 35-50%. BIS monitoring will be applied and level of anaesthetia will be titrated to keep a BIS value of 40-60. Intravenous remifentanil infusion between 0.1-0.25mcg/kg/min will be given and this will be titrated to optimal haemodynamic parameters. Muscle relaxants can be given during the operation as required.

Intravenous phenylephrine, ephedrine or fluid administration with colloid or crystalloid will be given at the discretion of the anaesthesiologist for management of hypotension. Hypertension or tachycardia will be managed by titrating the remifentanil infusion up to 0.25mcg/kg/min or sevoflurane up to 1.5 MAC. Intravenous anti hypertensive agents such as beta blockers (eg. esmolol, labetolol), hydralazine, glyceryl trinitrate, and phentolamine can be given if hypertension persists.

Thermal blanket will be used with the aim of keeping a core temperature of 35.5-37.5 degrees Celsius. Ondansetron 4mg IV can be given 30 minutes before end of surgery.

Sevoflurane and remifentanil infusion will be switched off at the end of the procedure. Reversal of muscle relaxation can be obtained if required with neostigmine 50mcg/kg IV and atropine 20mcg/kg IV after the operation. Patients will subsequently be transferred to the post anaesthetic care unit (PACU) for monitoring for at least 30 minutes.

Group P

Patients in group P will be anaesthetized according to the following protocol:

Monitoring and other anaesthetic procedures including the management of hypertension and hypotension will be the same as group S. The only difference is that induction and maintenance of general anaesthesia will be conducted using total intravenous infusion of propofol. Sevoflurane will not be used, and oxygen and air would be given to provide a FiO2 of 30-50%.

Target controlled infusion (TCI) with modified Marsh effect site model (Fresenius Kabi) will be used for induction and maintenance of general anaesthesia. Level of anaesthesia will be titrated to produce a BIS value of between 40-60. As with patients in group S, remifentanil will be infused at a rate of between 0.1-0.25mcg/kg/min.

Analgesic modalities and pain assessment

Both groups (Groups S and P)

Dental surgeon will provide local infiltration with 2.7ml of 2% lignocaine with 1:80,000 adrenaline around the base of the gum of each third molar tooth. Morphine sulphate at a bolus dose of 0.025-0.075 mg/kg will be given intravenously before skin incision.

Resting pain scores will be checked every 5 minutes in the post anaesthetic care unit. 2mg boluses of intravenous morphine sulphate will be given every 5 minutes until the NRS pain score is less than 4/10. Respiratory rate, oxygen saturation, Ramsay sedation scores, blood pressure and heart rate will be monitored every 5 minutes while the patient is in the post anaesthetic care unit.

When the patient resumes fluid diet on postoperative day 0, oral paracetamol 500mg q6h and oral dihydrocodeine 30mg q6h will be prescribed on an as needed basis when NRS pain score is more than 3/10 for three days. Both analgesics will be given together.

In the ward, pain related parameters like the numerical rating scales (NRS) pain scores at rest and mouth opening, and side effects will also be recorded every 1 hour for 6 hours, and then once every 4 hours. Patients will be given a diary to record NRS pain scores at rest and with mouth opening, analgesic consumption, and side effects at 24th, 48th and 72nd hour after operation. Global pain satisfaction using a scale of 0-10 (0 being least satisfied and 10 being most satisfied) will be recorded on postoperative day 3.

Monitoring of vital signs will be at the discretion of the attending dental surgeon once the patient returns to ward, and final hospital discharge will also be determined by the attending dental surgeon.

A brief home telephone interview will be conducted at 3 months to assess the incidence of chronic pain. The severity of pain, if present, would be recorded using NRS at rest and on mouth opening from 0-10.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III
* Age 18 to 80 years old
* Scheduled for elective extraction of impacted bilateral third molar teeth under general anaesthesia in Queen Mary hospital.

Exclusion Criteria:

* Known drug allergy to propofol, opioids, non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2 inhibitors, paracetamol.
* Alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120µmol/L
* Patients with liver dysfunction (Plasma bilirubin over 34 micromol/L, INR over 1.7, ALT and AST over 100U/L)
* Impaired or retarded mental state
* BMI > 35kg/m2
* History of chronic pain
* Pregnancy
* Local infection
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
pain score | up to postoperative day 3
  measure pain scores at rest and mouth opening using numeral rating scale

SECONDARY OUTCOMES:
analgesic consumption | up to postoperative day 3
  record analgesic consumption base on patient drug record
side effects of analgesics used | up to postoperative day 3
  pruritus, dizziness, nausea, vomiting, constipation etc.
intraoperative vital signs | during surgery
  blood pressure
intraoperative vital signs | during surgery
  heart rate
intraoperative vital signs | during surgery
  oxygen saturation
presence of persistent pain | 3 months after surgery
  presence of chronic pain after surgery (Yes or No), and severity of pain using NRS 0-10 if pain is present
severity of persistent pain | 3 months after surgery
  severity of pain using NRS 0-10 if pain is present

CONTACTS AND LOCATIONS:
Overall Officials: Stanley SC Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided